CLINICAL TRIAL: NCT06029868
Title: Improving the Process of Dryness, Limited Movement, and Joint Pain Using the Black Seed in Osteoarthritis: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Black Seed Oil in Treatment of Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsar international campus (Other)
Responsible Party: Principal Investigator, Mohammad Khodashenas Roudsari, Mohammad khodashenas roudsari ,Assistant prof of internal medicine, Ramsar international campus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.BUMS. REC.1398.020
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black seed (Experimental): Black seed oil capsule taken orally
  Interventions: Dietary Supplement: Black seed oil capsule
- Placebo (Placebo Comparator): Placebo capsule taken orally
  Interventions: Dietary Supplement: Placebo Black seed oil capsule

INTERVENTIONS:
Dietary Supplement: Black seed oil capsule — 700 mg black seed soft gel capsule once a day from Gorgan Essential Oil Pharmaceutical Company,
  Arms: Black seed
Dietary Supplement: Placebo Black seed oil capsule — Placebo Black seed oil capsule
  Arms: Placebo

SUMMARY:
Osteoarthritis is a continual illness of joints. We aim to investigate the effect of Nigella sativa oil in comparison with placebo on the reduction of osteoarthritis pain.

This study is a double-blinded, randomized, controlled trial study, conducting in Vali-e-Asr Hospital in 2019, in Birjand, on patients with mild osteoarthritis. The Western Ontario and McMaster Universities Osteoarthritis Index is applied to score the functional status of participants' joints.

DETAILED DESCRIPTION:
This study was a randomized controlled trial. Regarding to the inclusion criteria, 110 osteoarthritis patients were included in this study based on clinical signs, physical examination and radiological signs. In the next step, a fully explanation was given to the participants around the conditions of conducting the research, and then the informed consent were collected. Subsequently, patients were randomly divided into two groups of recipients; black seed soft gel capsules (intervention) and placebo equally in accordance with demographic information. Furthermore, the two groups were randomly classified regarding to age, consequently the study population was divided into subgroups of categorized ages. Thereafter, an equal number of each subgroup was randomly selected and divided into two groups to take black seed and placebo. Therefore, the two groups were similar, but the exact membership of individuals in the groups were random. Due to the higher prevalence of osteoarthritis among women in the community, the number of female cases were higher. It should be noted that the experimenters as well as patients did not know who was receiving a particular treatment (Double-blinded study). Prior to commencing the study, participants were asked to take a regular 48-day course of anti-inflammatory therapy. The cases in the intervention group took 700 mg of black seed soft gel capsule once a day from Gorgan Essential Oil Pharmaceutical Company, and the control group were treated by placebo capsules in the same-color and shape of the drug, with a taste of rice bran. Moreover, questionnaires were filled to record demographic information of both groups including age, sex, history medication and diet. The condition of participants were evaluated twice before the treatment and 48 days after the onset of black seed. At the end of each period, joint pain scores, the range of activity, and the dryness of the joints of all patients were assessed, and their mean were measured.

Data collection tools:

Scoring the functional status of individuals' joints were evaluated by applying Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)[2]. The WOMAC questionnaire was published in the 1908s to assess osteoarthritis of hip and knee, which is a standard criterion for assessing the health status of patients' self-reported activity. Three criteria should be measured ranging between zero to 4 for each question, by the end of each evaluation period: reduce pain is identified based on the mean for the first 5 WOMAC questions (from no pain to severe pain), the 6th and 7th questions were specified for joint dryness (from no dryness to severe limitation),and Joint movement is determined based on the average of questions 0 to 24 (from no problem to severe limit).

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral involvement of one or more joints for over 4 months,
* ability to walk
* ability to stay throughout the study period
* no history of underlying inflammatory disease (arthropathy / rheumatoid arthritis),
* absence of diabetes,
* no history of allergy to black seed
* absence of hyperuricemia (<338 umol/l) or history of gout,
* absence of recent injury and trauma to the joint with osteoarthritis,
* absence of intra articular injection of corticosteroids in the last 4 months,
* lack of sensitivity to NSAIDS,
* no underlying liver and kidney disease or history of peptic ulcer Or gastrointestinal bleeding, Congestive Heart Failure, hypertension, and hyperkalemia ,
* no fever
* absence of obvious Complete Blood Count disorders, coagulopathy, hematologic or neurological disorders ,
* no alcohol consumption

Exclusion Criteria:

* pregnancy,
* breast feeding,
* pregnancy-related decision
* obesity (BMI> 30 kg /m2).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Knee joint pain | 48 days
  Scoring the functional status of individuals' joints were evaluated by applying Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) .reduce pain is identified based on the mean for the first 5 WOMAC questions (from no pain to severe pain)
joint movement limitation | 48 days
  Scoring the functional status of individuals' joints were evaluated by applying Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Joint movement is determined based on the average of questions 0 to 24 (from no problem to severe limit).
joint dryness | 48 days
  Scoring the functional status of individuals' joints were evaluated by applying Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). the 6th and 7th questions were specified for joint dryness (from no dryness to severe limitation)

CONTACTS AND LOCATIONS:
Locations (1):
- Ramsar international campus, Ramsar, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: No